CLINICAL TRIAL: NCT01222429
Title: Practice-Based Nutrition Intervention
Brief Title: Practice Based Nutrition Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PBNI-1
Record Dates: First submitted 2010-10-12; First posted 2010-10-18 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Vegan

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- diet following American Diabetes Association guidelines (Active Comparator): Participants will follow diets based on ADA guidelines. This group will also receive weekly nutrition classes.
  Interventions: Other: diet following ADA guidelines
- vegan diet (Experimental): Participants in the intervention group will follow a low-fat, vegan diet for 20 weeks, and will attend nutrition classes in the form of a weekly support group.
  Interventions: Other: vegan diet

INTERVENTIONS:
Other: vegan diet — Intervention group participants will follow a low-fat vegan diet and will receive instruction on this diet through the course of the study
  Arms: vegan diet
Other: diet following ADA guidelines — participants will be given instruction on the ADA guidelines for diabetes, and will follow an individualized plan based on these guidelines
  Arms: diet following American Diabetes Association guidelines

SUMMARY:
This study aims to test a dietary intervention for diabetes in a medical practice setting, with the aim of developing a model for diabetes care that can be used widely. The investigators hypothesize that a low-fat vegan diet will be effective for management of diabetes and will be feasible in a practice-based setting.

DETAILED DESCRIPTION:
Specific Aim 1 tests the hypothesis that the nutrition intervention (low fat, low-GI vegan diet) improves glycemic control, body weight, plasma lipid concentrations, blood pressure, and indices of renal function in a within-group analysis.

Specific Aim 2 tests the hypothesis that the nutrition intervention (low fat, low-GI vegan diet) is more effective than standard nutrition care for improving glycemic control, body weight, plasma lipid concentrations, blood pressure, and indices of renal function in individuals with type 2 diabetes

Specific Aim 3 tests the hypothesis that a low-fat vegan diet is sustainable among individuals with type 2 diabetes for a 20-week period, with weekly classes, and in a follow-up period of one year with limited professional support.

Specific Aim 4 tests the hypothesis that a low-fat vegan diet has an acceptability that is comparable to that of standard nutrition care among individuals with type 2 diabetes.

Specific Aim 5 tests the hypothesis that the effects of the dietary interventions on A1c and body weight are reduced in individuals with the A1 allele of the Taq1A and Taq1B polymorphism

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of type 2 diabetes mellitus, as defined by a fasting plasma glucose concentration ≥126 mg/dl on 2 occasions or a prior physician's diagnosis of type 2 diabetes with the use of hypoglycemic medications for at least 6 months
2. male or female
3. A1c between 6.5% and 10.5%
4. age at least 18 years
5. ability and willingness to participate in all components of the study
6. willingness to be assigned to either a low-fat, vegan diet or to standard nutrition care
7. diabetes medications unchanged for 1 month prior to volunteering for the study
8. patient of Dr. Mark Sklar

Exclusion Criteria:

1. body mass index >45 kg/m2
2. alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
3. use of recreational drugs in the past 6 months (past drug use, if fully recovered, is not a criteria for exclusion)
4. pregnancy or plans to become pregnant
5. history of severe mental illness (with current unstable status)
6. likely to be disruptive in group sessions (as determined by research staff)
7. Signs/symptoms of acute uncontrolled diabetes (including but not limited to polyuria, polydipsia, blurred vision, uncontrolled weight loss)
8. unstable medical status
9. already following a low-fat, vegetarian diet
10. an inordinate fear of blood draws
11. inability to maintain current medication regimen
12. lack of English fluency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1C (diabetes management) | assessment at baseline (0 weeks)
hemoglobin A1C (diabetes management) | assessment at 10 weeks
hemoglobin A1C (diabetes management) | assessment at 20 weeks
hemoglobin A1C (diabetes management) | assessment at one-year follow-up
lipid profile (serum cholesterol--total, LDL, HDL; triglycerides) | assessment at baseline (0 weeks)
lipid profile (serum cholesterol--total, LDL, HDL; triglycerides) | assessment at 10 weeks
lipid profile (serum cholesterol--total, LDL, HDL; triglycerides) | assesment at 20 weeks
lipid profile (serum cholesterol--total, LDL, HDL; triglycerides) | assessment at one-year follow-up
body weight | assessment at baseline (0 weeks)
body weight | assessment at 10 weeks
body weight | assessment at 20 weeks
body weight | assessment at one-year follow-up
indices of renal function (serum creatinine, microalbumin) | assessment at baseline (0 weeks)
indices of renal function (serum creatinine, microalbumin) | assessment at 10 weeks
indices of renal function (serum creatinine, microalbumin) | assessment at 20 weeks
indices of renal function (serum creatinine, microalbumin) | assessment at one-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Barnard, MD, Principal Investigator — Washington Center for Clinical Research

REFERENCES:
- [Derived] Barnard ND, Levin SM, Gloede L, Flores R. Turning the Waiting Room into a Classroom: Weekly Classes Using a Vegan or a Portion-Controlled Eating Plan Improve Diabetes Control in a Randomized Translational Study. J Acad Nutr Diet. 2018 Jun;118(6):1072-1079. doi: 10.1016/j.jand.2017.11.017. Epub 2018 Feb 15. PMID 29398571